CLINICAL TRIAL: NCT00134251
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Ascending Dose, Parallel Group Study Exploring Effects of SLV308 up to 42 mg/Day Administered as an Adjunctive Therapy to L-Dopa in Patients With Advanced Stage Parkinson's Disease
Brief Title: Ascending Dose Tolerability/Safety of SLV308 for the Treatment of Parkinson's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S308.3.005; EuDract no 2005-002432-10
Record Dates: First submitted 2005-08-22; First posted 2005-08-24 (Estimated); Last update posted 2009-01-30 (Estimated); Status verified 2009-01

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; adjunctive to L-dopa therapy; Advanced stage Parkinson's disease
MeSH Terms: conditions — Parkinson Disease | interventions — pardoprunox

INTERVENTIONS:
Drug: SLV308

SUMMARY:
This study is a multicenter, randomized, double-blind, placebo controlled, parallel group study of a seven-week ascending dose period of SLV308 adjunctive to L-dopa treatment in patients with advanced stage Parkinson's disease (PD) and dose-dependent motor fluctuations. Patients (outpatients) will be randomized to one of three different treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have signed an informed consent; diagnosis of idiopathic PD.
* Presence of recognizable "on" and "off" stages
* Minimum hours of "off" time per day of 2.5 hours
* Able to keep diaries.

Exclusion Criteria:

* Unclear diagnosis or a suspicion of other parkinsonian syndromes
* Have undergone surgical treatment for PD
* History of non-response to L-dopa.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-10

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (10):
- Bulgaria (6):
  - Site 16, Plovdiv
  - Site 11, Sofia
  - Site 12, Sofia
  - Site 13, Sofia
  - Site 14, Sofia
  - Site 15, Sofia
- Site 21, Guardamangia, Malta
- Serbia (3):
  - Site 31, Belgrade
  - Site 34, Belgrade
  - Site 33, Niš